CLINICAL TRIAL: NCT05902871
Title: Direct Selective Laser Trabeculoplasty for Primary Open Angle Glaucoma and Ocular Hypertension and Normal Tension Glaucoma in Ethnic Chinese Population - The Zhuiguangzhe Trial
Brief Title: Direct Selective Laser Trabeculoplasty in Ethnic Chinese Population
Acronym: Zhuiguangzhe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BelkinVision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: #China-2022-01 (CA-PL-01-008)
Record Dates: First submitted 2023-05-10; First posted 2023-06-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension; Normal Tension Glaucoma
Keywords: Glaucoma; High intraocular eye pressure; Normal tension open angle glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Low Tension Glaucoma; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSLT with Eagle (Group 1) (Experimental): Single treatment 360 degrees with laser energy of 1.2 mJ
  Interventions: Device: External Automatic Glaucoma Laser; Procedure: Direct Selective Laser Trabeculoplasty
- DSLT with Eagle (Group 2) (Experimental): Single treatment 360 degrees with laser energy of 1.8 mJ
  Interventions: Device: External Automatic Glaucoma Laser; Procedure: Direct Selective Laser Trabeculoplasty

INTERVENTIONS:
Device: External Automatic Glaucoma Laser — Trans-limbal, direct selective laser trabeculoplasty (DSLT) instrument that directs laser energy through the sclera around the limbus overlying the trabecular meshwork and treats 360 degrees of the angle is treated simultaneously
  Other Names: Eagle
Procedure: Direct Selective Laser Trabeculoplasty — Surgical procedure that utilizes a laser to improve fluid drainage in the eye and reduce intraocular pressure
  Other Names: DSLT

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Direct Selective Laser Trabeculoplasty (DSLT) in ethnic Chinese participants with Primary Open Angle Glaucoma (POAG), Ocular Hypertension (OHT), or Normal Tension Glaucoma (NTG).

DETAILED DESCRIPTION:
After informed consent is obtained, potential study participants will undergo a hypotensive medication washout period as applicable. Patients will then be re-assessed for eligibility and treated with DSLT if they meet the inclusion/exclusion criteria. The first 5 patients will be treated 360 degrees with laser energy of 1.2 millijoule (mJ) (Group 1). If all 5 Group 1 patients pass the pre-defined safety endpoint at Week 1, then the next 40 patients will be treated 360 degrees with laser energy of 1.8 mJ (Group 2). Patients will attend one treatment visit and up to 9 follow-up visits, remotely or at the clinic. Individual duration of participation is approximately 12 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Chinese ethnicity with corrected visual acuity greater than 6/18 in both eyes.
* Diagnosed with mild to moderate primary open angle glaucoma, ocular hypertension, or normal tension open angle glaucoma.
* Willing and able to participate in a 12-month study, comply with the study procedures, and adhere to the follow-up schedule.
* Capable of giving informed consent.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Eye conditions as specified in the protocol.
* Use of medications as specified in the protocol.
* Unable to provide a reliable visual field test.
* Women who are pregnant or may become pregnant during the study.
* Prior surgery in the study eye.
* In a vision-dependent profession such as pilot or commercial driver.
* Other protocol-specified exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in IOP at Month 6 | Baseline (Day -7 to 0) (post washout and pretreatment), Month 6
  Intraocular pressure (IOP) will be assessed with Goldmann applanation tonometry and recorded in millimeters mercury (mmHg). Change from baseline is defined as the difference between baseline (washed out for medicated patients) IOP and (washed out for medicated patients) IOP measured at Month 6 for each participant enrolled in the study. A negative change from baseline will represent an improvement.

SECONDARY OUTCOMES:
Mean Percent Reduction from Baseline in IOP at Month 6 and Month 12 | Baseline (Day -7 to 0) (post washout and pretreatment), Month 6, Month 12
  Intraocular pressure (IOP) will be assessed with Goldmann applanation tonometry and recorded in millimeters mercury (mmHg). Change from baseline is defined as the difference between baseline (washed out for medicated patients) IOP and (washed out for medicated patients) IOP measured at the respective timepoints (Month 6 and Month 12). A positive percent reduction will represent an improvement.
Proportion of Subjects with at least 20 percent reduction in IOP from Baseline in IOP for POAG and OHT and at least 15 percent reduction in IOP for NTG at Month 6 with no Secondary Surgical Intervention (SSI) or Inability to Washout | Baseline (Day -7 to 0) (post washout and pretreatment), Month 6, Month 12
  Intraocular pressure (IOP) will be assessed with Goldmann applanation tonometry and recorded in millimeters mercury (mmHg). A secondary surgical intervention (SSI) is defined as a procedure in addition to DSLT that is conducted to manage/lower IOP. A higher proportion with the specified reduction will represent an improvement.
Change from Baseline in Number of Glaucoma Medications at Month 6 and Month 12 | Screening (Day -45 to -1) (prewashout and pretreatment)/Visit 1 (Day 0) (pretreatment), Month 6, Month 12
  The number of glaucoma-related medications in use will be recorded. For medicated subjects, the Screening visit is considered baseline. For naïve (unmedicated) subjects, Visit 1 is considered baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Raz Prag, Study Director — Alcon Research, LLC
Locations (2):
- C-Mer Eye Clinic, Hong Kong, China
- SERI, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No